CLINICAL TRIAL: NCT03773809
Title: Impact of Vitamin D3 Administration on Cardiac Autonomic Tone in Asthma COPD Overlap(ACO) Patients: A Blinded Randomized Control Trial
Brief Title: Impact of Vitamin D3 Administration on Cardiac Autonomic Tone in Asthma Chronic Obstructive Pulmonary Disease(COPD) Overlap Patients
Acronym: COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Salsa Bil Nahar, Resident, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: No. BSMMU/2018/478
Record Dates: First submitted 2018-11-29; First posted 2018-12-12 (Actual); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Asthma-COPD Overlap Syndrome; Vitamin D Deficiency; Cardiac Autonomic Tone
Keywords: ACO; HRV; Vitamin D deficiency
MeSH Terms: conditions — Asthma-Chronic Obstructive Pulmonary Disease Overlap Syndrome; Vitamin D Deficiency | interventions — Vitamin D

STUDY DESIGN:
Intervention Model Description: Baseline group:
  This group will include 60 vitamin D3 deficient ACO patients.
  Group A:
  Group A0: Vitamin D3 deficient ACO patients with placebo at day 0. Group A90: Vitamin D3 deficient ACO patients with placebo at day 90
  Group B:
  Group B0: Vitamin D3 deficient ACO patients with vitamin D3 at day 0. Group B90: Vitamin D3 deficient ACO patients with vitamin D3 at day 90.
  All the patients will be similar by age, sex and BMI
Who Masked: Participant, Investigator
Masking Description: Both the patients and the principal investigator will remain blind to the intervention given. After the end of follow up, at the time of data analysis principal investigator will be provided with the information about which patient isgoven placebo and which patient isgivev drug.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A0 (Placebo Comparator): Vitamin D3 deficient ACO patients with placebo at day 0.
  Interventions: Other: placebo
- Group A90 (Placebo Comparator): Vitamin D3 deficient ACO patients with placebo at day 90.
  Interventions: Other: placebo
- Group B0 (Active Comparator): Vitamin D3 deficient ACO patients with vitamin D3 at day 0.
  Interventions: Other: Vitamin D capsule
- Group B90 (Active Comparator): Vitamin D3 deficient ACO patients with vitamin D3 at day 90.
  Interventions: Other: Vitamin D capsule

INTERVENTIONS:
Other: Vitamin D capsule — The intervention was given by oral administration of vitamin D3 capsule each of which contains 40000 IU of vitamin D3. The capsule was manufactured and supplied by Beximco Pharmaceutical Limited, Bangladesh. The placebo was also be manufactured and supplied by the same pharmaceutical company and was similar in size shape & appearance to vitamin D3 capsule but contained all the ingredients of vitamin D capsule other than the vitamin D3
  Other Names: oral administration of Vitamin D capsule
  Arms: Group B0; Group B90
Other: placebo — oral administration of placebo
  Arms: Group A0; Group A90

SUMMARY:
Title:Impact of vitamin D administration on cardiac autonomic tone in Asthma Chronic Obstructive Pulmonary Disease (COPD) Overlap patients: A blinded randomized control trial.

Background: Respiratory disease is closely associated with cardiovascular disease. Reduced Heart Rate Variability (HRV), reflecting impaired autonomic activity have been reported in both asthma and COPD. Vitamin D deficiency is a common feature in Asthma COPD Overlap (ACO) patient. Relationship between vitamin D deficiency and low HRV has been reported. Vitamin D administration has been reported to improve cardiac autonomic modulation in healthy subjects in response to external stressor. Objective: To assess the changes in cardiac autonomic tone after vitamin D administration for 90 days in vitamin D deficient ACO patients.

Hypothesis:Null: Vitamin D administration does not have impact on cardiac autonomic tone in vitamin D3 deficient ACO patient.

.Method: This randomized controlled trial will be conducted by Department of Physiology, Bangabandhu Sheikh Mujib Medical University (BSMMU), Shahbag, Dhaka from September' 2017 to August' 2018. For this study, a total number of 60 subjects (age > 40 years, both male and female) will be randomly selected. 30 diagnosed vitamin D deficient Asthma COPD Overlap (ACO) patients will form group A and another 30 diagnosed vitamin D3 deficient ACO patients with similar age, sex, (Body Mass Index) BMI will constitute control group B. Patients of study group B0 will take vitamin D3 with a prescribed schedule for 3 months and followed up after 3 months (group B90). On the other hand patients of group A1 will be given placebo and followed up after 3 months (group A90). All these patients will continue their medication prescribed by physician during these 3 months. On the basis of data recording - group B1 and group B90 will constitute pre and post vitamin D group whereas group A0 and group A90 will represent pre and post placebo follow up at day 0 and day 90. Cardiac autonomic nerve function will be assessed by recording ECG & Heart Rate Variability (HRV) analysis by a data acquisition device, powerlab 8/35, AD instruments, Australia. HRV measures of all patients will be recorded at baseline.Then after 3 months of follow up it will be recorded in both groups at day 90. Serum 25(OH)D level will be measured of all subject at day 0 and day 90. For statistical analysis unpaired and paired "t" test will be done by using Microsoft Office Excel Word version 2016

DETAILED DESCRIPTION:
Previous studies reported earlier age of onset, symptom with longer duration, more exacerbation and devoid of adequate health care in Asthma Chronic Obstructive Pulmonary Disease (COPD) Overlap (ACO) patients compared to asthma and Chronic Obstructive Pulmonary Disease (COPD) alone. However their prevalence rate was reported between 15 and 55%. Existence of asthma and COPD has been reported in between 15-20% of patient. There is no population based data on ACO patients in Bangladesh. But one study very recently reported 11.6% of Asthma COPD Overlap (ACO) patients in this country. Thus it is of utmost importance to perform more research on this significant disease.

Several studies investigated autonomic function in asthma and COPD patients. Both asthma and COPD affect cardiac autonomic function. Poor asthma control is associated with lower HRV, depressed sympathetic and enhanced parasympathetic modulation. It has reported that the risk of cardiovascular disease in COPD is increase by 2 to 3 fold and it is the leading cause of death in mild to moderate COPD. But to the best of our knowledge no study investigated the cardiac autonomic function of ACO patients.

Vitamin D deficiency is a common feature in ACO patient. Previous studies demonstrated the relationship between vitamin D deficiency and reduced HRV resulting in incidence of cardiovascular disease. Only one study reported the effect of vitamin D administration on HRV. They enrolled young healthy subjects and observed the effect of vitamin D on HRV in response to physiological stressor such as angiotensin II induced stress. All these subjects were vitamin D insufficient and their result showed improvement of sympathovagal balance after administration of vitamin D. With this experimental observation we can expect, administration of vitamin D in vitamin deficient ACO patients might improve cardiac autonomic function and thereby protect them from the risk cardiovascular morbidity and mortality.

However vitamin D appears to be a simple, cost effective treatment to reduce cardiovascular disease associated risk by improving function of autonomic nerve function in both healthy and chronic disease population worldwide. But the volume of information regarding the effect of vitamin D administration in ACO patients is not enough for reaching any final conclusion. Moreover, with the best of our knowledge no study have been conducted to observe the effects of this fat soluble vitamin on HRV in vitamin D deficient, stable patients with ACO.

Therefore, on the basis of this background the present study has been designed to evaluate the effects of Vitamin D on heart rate variability in D deficient, stable patients with ACO. This study will draw attention of the physicians on the cardiac autonomic status of ACO patients and the effects of Vitamin D on it.

General Objectives:

This study will assess the impact of vitamin D therapy on cardiac autonomic tone in vitamin D deficient ACO patients by heart rate variability analysis.

Specific Objectives:

* To measure HRV by time domain and frequency domain and nonlinear methods in vitamin D deficient ACO patient at baseline.
* To measure all these above parameters after 3 months of vitamin D and placebo administration.
* To Compare pre and post intervention HRV parameters in both vitamin D group and placebo group of ACO patients.

Methods

1. Study design:

   This study will be a randomized controlled trial where experiment will be done with either vitamin D therapy or with placebo for 3 months onward.
2. Study center:

   This study will be carried out in the department of Physiology of Bangabandhu Sheikh Mujib Medical University (BSMMU), Dhaka under continuous supervision and monitoring.
3. Period of study:

   This study will commence from September, 2017 and expected to end by August, 2018.
4. Ethical Clearance:

   The protocol of this study involving the human subjects will be submitted to Institutional Review Board (IRB) of Bangabandhu Sheikh Mujib Medical University (BSMMU) for ethical and other technical approval before commencing the actual study.this project is a part of an ongoing research which was approved by Institutional Review Board (IRB) of Bangabandhu Sheikh Mujib Medical University (BSMMU).
5. Sampling:

Sample size:

Total 60 subjects will be recruited in this study, which is designed for randomized controlled trial on the basis of outcome measures (effect size) i.e. estimation of mean differences between pre & post intervention mean of the study which has already been published in a cross sectional study that assess the association of vitamin D deficiency with cardiac autonomic activity. Sample size based on effect size .

Sampling Technique:

Simple random sampling will be adopted to select the patients. According to the selection criteria total 60 subjects of both male and female with specific age range suitable for the aim and objective of the study will be enrolled. These diagnosed ACO patients (diagnosed by applying the "tick box" approach recommended by the joint committee of GOLD & GINA from Out Patient Department (OPD) of NIDCH) will be selected by clinicians in OPD of National Institute of the Disease of Chest and Hospital (NIDCH).

Grouping of the subjects:

After a careful brief interview, selection and enrollment of the subjects for this study will be done. All the subjects will be divided into following groups according to the objectives of the study

Baseline group:

This group will include 60 vitamin D deficient ACO patients.

Group A:

25 diagnosed vitamin D deficient ACO patients will be included in this group and they will be given vitamin D. This group will be further divided into the following group.

Group A0: Vitamin D deficient ACO patients with placebo at day 0. Group A90: Vitamin D deficient ACO patients with placebo at day 90

Group B:

25 diagnosed vitamin D deficient ACO patients will be included in this group and they will be given placebo. This group will be further divided into the following group.

Group B0: Vitamin D deficient ACO patients with vitamin D at day 0. Group B90: Vitamin D deficient ACO patients with vitamin D at day 90.

All the patients will be similar by age, sex and BMI.

8. Study intervention:

The intervention will be given by oral administration of vitamin D3 capsule each of which contain 40000 International Unit (IU) of vitamin D. The capsule will be manufactured and supplied by Beximco Pharmaceutical Limited, Bangladesh. The placebo will also be manufactured and supplied by the same pharmaceutical company and will be similar in size shape & appearance to vitamin D capsule but it will contain sucrose powder. All patients will be advised to take 2 capsule after breakfast on a fixed day of the week for 3 consecutive months.

At the time of enrollment all patients will be randomized to one of the two interventions (placebo or vitamin D) immediately. The intervention will be double blind randomized and cross over design so that each patient will act as his/her control. Each participant of the placebo group & vitamin D3 group will be studied before & after intervention and comparison will be done between these two groups. In addition comparison will be done post intervention data of placebo & vitamin D group.

9. Study procedure:

On the first day of enrollment the researcher will introduce herself to the patient and ask for permission to talk to them. Then she will cordially explain about the objectives, purpose, and procedure of the study on the day of enrollment. The benefit as well as risk (if any) of the study should be carefully mentioned. Special emphasis will be given on explaining how he/she will be benefited from this study. The patient will be motivated for voluntary participation and will be allowed to withdraw him or herself from the study even after participation, whenever the patient feels uneasy. If he or she agrees to be a part of the study, an informed written consent will be taken in a prescribed form. Detailed family history, medical history and thorough physical examination of each patient will be done and all the information will be recorded in a standard data sheet. Then all the patients will be requested to attend the Department of Physiology at 8:30 am on the day of biochemical examination On the examination day, 5 ml of venous blood will be collected and taken to the biochemistry laboratory as soon as possible for the estimation of serum 25(OH)D. BMI will also be calculated by recording height weight. After getting the biochemical report, the final selection will be done, according to the inclusion and exclusion criteria..

Randomization and blinding: As it is not possible to exclude ACO patient with hypertension and/or diabetes , we will apply stratified randomization technique according to these two confounding factors. Four strata will be formed, as hypertension, diabetes, diabetes with hypertension and without hypertension and diabetes. Whenever a patient will be selected for enrollment, he will be given an Identification Number (ID) and assigned to one of the four strata according to his characteristics.

The randomization and blinding design was developed by a faculty of the Department of Physiology who is not included in the study team. The ID number and stratification will informed to the faculty. She (the faculty) will then then randomly allocate the patient in either group A (placebo) or group B (vitamin D) considering his strata so that both the group had equal number of patients from each strata. The faculty will then note down the patient ID in the allotted group and supplied principal investigator (PI) the drug (placebo or vitamin D) according to the allotted group.

At the end of the study, the faculty will provide the list of the patient's ID with allotted group to the PI

Data collection: All the selected patients will be then requested to come to the Department again on the next day for the HRV test with proper preparation.

Preparation for HRV test: Preparation for the test will be explained to them. For HRV examination, the subject will have to take their meal by 9:00 pm and need to have a sound sleep in the previous night. From previous night up to the time of examination, they will be requested not to undergo any physical or mental stress and also avoid taking any sedatives or any other drugs that affect central nervous system (Task force, 1996).The patients will be requested to take light breakfast in the morning without tea or coffee. After that, the selected subjects will be kept in complete bed rest in supine position for 10-15 minutes in the cool and calm laboratory environment to adjust with the lab conditions. During this period, the subject will be advised not to talk, eat or drink and also not to perform physical or mental activity even sleep .

Laboratory conditions and recording of HRV: The recording of HRV measures will be done by 8 active channels, power lab 8/35 (AD instrument, Australia), in the Autonomic Nerve Function Laboratory of Department of Physiology, BSMMU. The temperature of the laboratory will be maintained at 25°C-28°C and lights will be kept dim. It will also be maintained noise free. Door of the lab will be closed and no one will be allowed to enter the room during the test except the investigator and the subject.

Once the HRV recording will be completed, the patients will be provided the drug (containing placebo or vitamin D3 ) and will be asked to take 2 capsule per week for consecutive 90 days. The schedule of the therapy will be explained meticulously in detail to the patients. He/she will also be informed about the possible side effect of the drug (e.g. diarrhea). If the subject is able to understand everything explained to him, then he/she will be advised to continue the drug therapy for the consecutive 90 days. If the subject finds it difficult to understand the intervention or if any side effect of the drug appears, he/she will be asked to come to the department or to contact via telephone. During this period, the subjects will be regularly monitored and encouraged to be the part of this study by maintaining regular communication through telephonic calls several times a week. A good rapport will be built up to take time to time follow-up over telephone and visiting patient's place. In addition, scheduled appointment, hot-line and follow up will be maintained properly. If the subject finds it difficult to understand the intervention or if any side effect of the drug appears, he/she will be asked to come to the department or to contact via telephone. All the selected ACO patients will be allowed to continue standard therapeutic treatment as prescribed by the physician for these three months. Along with this, all the subjects of both the groups will be advised to continue a diet according to their own choice. Subsequently, all subjects will be requested to attend the Department of Physiology, BSMMU again on the 90th day for assessment of all the above-mentioned study variables. Any subject who fails to follow the study procedure exactly during the study period will be dropped and a new one will be included to fulfill the desired total sample size. At the end of the study i.e. after 90 day vitamin D3 will be given to all the patients of placebo group.

ELIGIBILITY:
Inclusion Criteria:

* • 40-80 years of age

  * Male
  * Middle class of socioeconomic condition:.
  * Stable patients of Asthma COPD Overlap (ACO) with >4 years of disease duration.
  * Vitamin D deficient (Serum 25-hydroxycholecalciferol, 25(OH)D level < 30 ng/ml).
  * Normal serum Ca+and inorganic phosphate level.
  * Hypertension with ACO.
  * Diabetes with ACO

Exclusion Criteria:

* Unstable patients with ACO (patients with exacerbation and medication changes in the past 30 days)
* With acute exacerbation of any pulmonary diseases, such as,

  * Bronchial asthma
  * Acute respiratory tract infection
  * Current tuberculosis
  * Pleural effusion
  * Emphysematous bullae
  * Interstitial lung disease
  * Pneumonectomy or pulmonary lobectomy
  * Pulmonary fibrosis.
* With acute exacerbation of any cardiac disease, like -

  * Unstable angina pectoris
  * Congestive heart failure
  * Myocardial infarction
  * Cardiac arrhythmia
* Rheumatoid arthritis.
* Inflammatory bowel disease.
* Chronic Renal Failure.
* Systemic lupus erythromatosIs.
* Musculoskeletal diseases.
* Any malignancy
* Systemic hypertension
* Use of drugs known to affect Central Nervous System (CNS) and vitamin D metabolism within 1 month prior to study, as,

  * Antiepileptics (Phenytoin, Carbamazepine)
  * Antibiotics (Clotrimazole, Rifampicin)
  * Antihypertensives (Nifedipine, Spironolactone)
  * Antiretroviral drugs (Ritononavir, Saquinavir)
  * Endocrine drugs (Cyproterone acetate)
  * Glucocorticoids
  * Bisphosphonate
  * Calcium supplement

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — male
Enrollment: 50 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
vitamin D concentration | Change from Baseline Serum vitamin D level at 90 days
  serum vitamin D level was measured at day 0 and after 90 days of vitamin D and placebo administration in vitamin D and in placebo group respectively
Mean R-R interval in milliseconds | Change from Baseline Mean R-R interval at 90 days
  Mean R-R interval was measured at day 0 and after 90 days of vitamin D and placebo administration in vitamin D and in placebo group respectively
Mean Heart Rate in beats/min | Change from Baseline Mean Heart Rate at 90 days
  Mean Heart Rate was measured at day 0 and after 90 days of vitamin D and placebo administration in vitamin D and in placebo group respectively
Standard deviation of RR interval (SDRR) in milliseconds | Change from Baseline Standard deviation of RR interval (SDRR) at 90 days
  Standard deviation of RR interval (SDRR) was measured at day 0 and after 90 days of vitamin D and placebo administration in vitamin D and in placebo group respectively
Coefficient of variation of all the R-R interval (CVRR) | Change from Baseline Coefficient of variation of all the R-R interval (CVRR) at 90 days
  Coefficient of variation of all the R-R interval (CVRR) was measured at day 0 and after 90 days of vitamin D and placebo administration in vitamin D and in placebo group respectively
Square root of the mean squared differences of successive RR interval (RMSSD) in milliseconds | Change from Baseline Square root of the mean squared differences of successive RR interval (RMSSD) at 90 days
  Square root of the mean squared differences of successive RR interval (RMSSD) was measured at day 0 and after 90 days of vitamin D and placebo administration in vitamin D and in placebo group respectively
Standard deviation of successive RR interval differences between adjacent RR intervals (SDSD) in milliseconds | Change from Baseline Standard deviation of successive RR interval differences between adjacent RR intervals (SDSD) at 90 dayss
  Standard deviation of successive RR interval differences between adjacent RR intervals (SDSD) was measured at day 0 and after 90 days of vitamin D and placebo administration in vitamin D and in placebo group respectively
Number of RR interval differing by >50 milliseconds from adjacent intervals divided by the total number of all RR intervals (pRR50%) in % | Change from Baseline Number of RR interval differing by >50 milliseconds from adjacent intervals divided by the total number of all RR intervals (pRR50%) at 90 days
  Number of RR interval differing by >50 milliseconds from adjacent intervals divided by the total number of all RR intervals (pRR50%) was measured at day 0 and after 90 days of vitamin D and placebo administration in vitamin D and in placebo group respectively
Total power (absolute) in frequency domain parameters of heart rate variability | Change from Baseline Total power (absolute) in frequency domain parameters of heart rate variability at 90 months
  Total power (absolute) in frequency domain parameters of heart rate variability was measured at day 0 and after 90 days of vitamin D and placebo administration in vitamin D and in placebo group respectively
Low Frequency (LF) power (absolute) in frequency domain parameters of heart rate variability | Change from Baseline Low Frequency (LF) power (absolute) in frequency domain parameters of heart rate variability at 90 days
  Low Frequency (LF) power (absolute) in frequency domain parameters of heart rate variability was measured at day 0 and after 90 days of vitamin D and placebo administration in vitamin D and in placebo group respectively
High Frequency (HF) power (absolute) in frequency domain parameters of heart rate variability | Change from Baseline High Frequency (HF) power (absolute) in frequency domain parameters of heart rate variability at 90days
  High Frequency (HF) power (absolute) in frequency domain parameters of heart rate variability was measured at day 0 and after 90 days of vitamin D and placebo administration in vitamin D and in placebo group respectively
Low Frequency (LF) power in normalised units (n.u) in frequency domain parameters of heart rate variability | Change from Baseline Low Frequency (LF) power in normalised units (n.u) in frequency domain parameters of heart rate variability at 90 days
  Low Frequency (LF) power in normalised units (n.u) in frequency domain parameters of heart rate variability was measured at day 0 and after 90 days of vitamin D and placebo administration in vitamin D and in placebo group respectively
High Frequency (HF) power in normalised units (n.u) in frequency domain parameters of heart rate variability | Change from Baseline High Frequency (HF) power in normalised units (n.u) in frequency domain parameters of heart rate variability at 90 days
  High Frequency (HF) power in normalised units (n.u) in frequency domain parameters of heart rate variability was measured at day 0 and after 90 days of vitamin D and placebo administration in vitamin D and in placebo group respectively
Ratio of Low frequency to High Frequency (HF) power in frequency domain parameters of heart rate variability | Change from Baseline Ratio of Low frequency to High Frequency (HF) power in frequency domain parameters of heart rate variability at 90 days
  Ratio of Low frequency to High Frequency (HF) power in frequency domain parameters of heart rate variability was measured at day 0 and after 90 days of vitamin D and placebo administration in vitamin D and in placebo group respectively

CONTACTS AND LOCATIONS:
Overall Officials: SULTANA FERDOUSI, FERDOUSI, Study Director — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (1):
- Dr Sultana Ferdousi, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Visweswaran RK, Lekha H. Extraskeletal effects and manifestations of Vitamin D deficiency. Indian J Endocrinol Metab. 2013 Jul;17(4):602-10. doi: 10.4103/2230-8210.113750. PMID 23961475
- [Background] Vinik AI, Maser RE, Mitchell BD, Freeman R. Diabetic autonomic neuropathy. Diabetes Care. 2003 May;26(5):1553-79. doi: 10.2337/diacare.26.5.1553. PMID 12716821
- [Background] Shaffer F, McCraty R, Zerr CL. A healthy heart is not a metronome: an integrative review of the heart's anatomy and heart rate variability. Front Psychol. 2014 Sep 30;5:1040. doi: 10.3389/fpsyg.2014.01040. eCollection 2014. PMID 25324790
- [Background] Heart rate variability: standards of measurement, physiological interpretation and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Circulation. 1996 Mar 1;93(5):1043-65. No abstract available. PMID 8598068
- [Background] Holick MF, Binkley NC, Bischoff-Ferrari HA, Gordon CM, Hanley DA, Heaney RP, Murad MH, Weaver CM; Endocrine Society. Evaluation, treatment, and prevention of vitamin D deficiency: an Endocrine Society clinical practice guideline. J Clin Endocrinol Metab. 2011 Jul;96(7):1911-30. doi: 10.1210/jc.2011-0385. Epub 2011 Jun 6. PMID 21646368
- [Background] Global Initiative for Asthma. Global Strategy for Asthma Management and Prevention, [Internet]. c2018. GOLD [updated 201; cited 2018 March 12] Available from: www.ginasthma.org
- [Background] Global Initiative for Asthma and Global Initiative for Chronic Obstructive Lung Disease. Diagnosis of Diseases of Chronic Airflow Limitation: Asthma, COPD and Asthma-COPD Overlap (ACO) [Internet]. A joint project of GINA and GOLD [updated April 2017; Cited 2017 Nov 12]. Available from: www.msc.es/organizacion/sns/plan CalidadSNS/pdf/GOLD_ACOS_2017.pdf
- [Result] Zupanic E, Zivanovic I, Kalisnik JM, Avbelj V, Lainscak M. The effect of 4-week rehabilitation on heart rate variability and QTc interval in patients with chronic obstructive pulmonary disease. COPD. 2014 Dec;11(6):659-69. doi: 10.3109/15412555.2014.898046. Epub 2014 Apr 30. PMID 24787632
- [Result] Wang TJ, Pencina MJ, Booth SL, Jacques PF, Ingelsson E, Lanier K, Benjamin EJ, D'Agostino RB, Wolf M, Vasan RS. Vitamin D deficiency and risk of cardiovascular disease. Circulation. 2008 Jan 29;117(4):503-11. doi: 10.1161/CIRCULATIONAHA.107.706127. Epub 2008 Jan 7. PMID 18180395
- [Result] Wang L, Song Y, Manson JE, Pilz S, Marz W, Michaelsson K, Lundqvist A, Jassal SK, Barrett-Connor E, Zhang C, Eaton CB, May HT, Anderson JL, Sesso HD. Circulating 25-hydroxy-vitamin D and risk of cardiovascular disease: a meta-analysis of prospective studies. Circ Cardiovasc Qual Outcomes. 2012 Nov;5(6):819-29. doi: 10.1161/CIRCOUTCOMES.112.967604. Epub 2012 Nov 13. PMID 23149428
- [Result] Voss A, Schulz S, Schroeder R, Baumert M, Caminal P. Methods derived from nonlinear dynamics for analysing heart rate variability. Philos Trans A Math Phys Eng Sci. 2009 Jan 28;367(1887):277-96. doi: 10.1098/rsta.2008.0232. PMID 18977726
- [Result] Vitamin D council. I tested my vitamin D level. What do my result mean? 2017 [Internet]. [Cited 2017 Oct 25]. Available from: https://www.vitamindcouncil.org/i-tested-my-vitamin-d-levelwhat-do-result-mean/
- [Result] Odler B, Ivancso I, Somogyi V, Benke K, Tamasi L, Galffy G, Szalay B, Muller V. Vitamin D deficiency is associated with impaired disease control in asthma-COPD overlap syndrome patients. Int J Chron Obstruct Pulmon Dis. 2015 Sep 24;10:2017-25. doi: 10.2147/COPD.S91654. eCollection 2015. PMID 26451099
- [Result] Nalbant A, Vatan MB, Varim P, Varim C, Kaya T, Tamer A. Does Vitamin D Deficiency Effect Heart Rate Variability in Low Cardiovascular Risk Population? Open Access Maced J Med Sci. 2017 Mar 22;5(2):197-200. doi: 10.3889/oamjms.2017.041. eCollection 2017 Apr 15. PMID 28507628
- [Result] Mann MC, Hollenberg MD, Hanley DA, Ahmed SB. Vitamin D, the autonomic nervous system, and cardiovascular risk. Physiol Rep. 2015 Apr;3(4):e12349. doi: 10.14814/phy2.12349. No abstract available. PMID 25902783
- [Result] Mann MC, Exner DV, Hemmelgarn BR, Turin TC, Sola DY, Ellis L, Ahmed SB. Vitamin D supplementation is associated with improved modulation of cardiac autonomic tone in healthy humans. Int J Cardiol. 2014 Mar 15;172(2):506-8. doi: 10.1016/j.ijcard.2014.01.058. Epub 2014 Jan 23. No abstract available. PMID 24502876
- [Result] Lutfi MF. Autonomic modulations in patients with bronchial asthma based on short-term heart rate variability. Lung India. 2012 Jul;29(3):254-8. doi: 10.4103/0970-2113.99111. PMID 22919165
- [Result] Hsu CH, Tsai MY, Huang GS, Lin TC, Chen KP, Ho ST, Shyu LY, Li CY. Poincare plot indexes of heart rate variability detect dynamic autonomic modulation during general anesthesia induction. Acta Anaesthesiol Taiwan. 2012 Mar;50(1):12-8. doi: 10.1016/j.aat.2012.03.002. Epub 2012 Apr 3. PMID 22500908
- [Result] Habib GMM, Nahar K, Habib F. Prevalence of Asthma and COPD Overlapping Syndrome (ACOS) in a busy primary care setting of Bangladesh. 1st IPCRG South Asian Scientific Conference: 2017 3-5 Agaust; Colombo. sri Lanka
- [Result] DeLuca GC, Kimball SM, Kolasinski J, Ramagopalan SV, Ebers GC. Review: the role of vitamin D in nervous system health and disease. Neuropathol Appl Neurobiol. 2013 Aug;39(5):458-84. doi: 10.1111/nan.12020. PMID 23336971
- [Result] Burt MG, Mangelsdorf BL, Stranks SN, Mangoni AA. Relationship between Vitamin D Status and Autonomic Nervous System Activity. Nutrients. 2016 Sep 13;8(9):565. doi: 10.3390/nu8090565. PMID 27649235
- [Result] Brzostek D, Kokot M. Asthma-chronic obstructive pulmonary disease overlap syndrome in Poland. Findings of an epidemiological study. Postepy Dermatol Alergol. 2014 Dec;31(6):372-9. doi: 10.5114/pdia.2014.47120. Epub 2014 Dec 3. PMID 25610352
- [Result] Bai JW, Mao B, Yang WL, Liang S, Lu HW, Xu JF. Asthma-COPD overlap syndrome showed more exacerbations however lower mortality than COPD. QJM. 2017 Jul 1;110(7):431-436. doi: 10.1093/qjmed/hcx005. PMID 28100824
- [Result] Akselrod S, Gordon D, Ubel FA, Shannon DC, Berger AC, Cohen RJ. Power spectrum analysis of heart rate fluctuation: a quantitative probe of beat-to-beat cardiovascular control. Science. 1981 Jul 10;213(4504):220-2. doi: 10.1126/science.6166045.